CLINICAL TRIAL: NCT05464823
Title: Feasibility of Combined Genomics/Transcriptomics for Patients With Lymphoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-0396; NCI-2022-05783 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2022-07-12; First posted 2022-07-19 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Molecular Testing (Other): Molecular Functional (MF) Portrait (a commercial test conducted by the sponsor of this study, BostonGene) in guiding lymphoma care.
  Interventions: Other: Molecular Functional Portrait

INTERVENTIONS:
Other: Molecular Functional Portrait — Participants will be asked to allow previously-collected tumor tissue to be used for the MF Portrait test

SUMMARY:
To learn more about the usefulness of molecular testing with the Molecular Functional (MF) Portrait (a commercial test conducted by the sponsor of this study, BostonGene) in guiding lymphoma care.

DETAILED DESCRIPTION:
Primary Objective:

• To determine the feasibility and turnaround of clinical WES and transcriptome sequencing

Secondary Objectives:

* To determine the frequency of actionable DNA and RNA alterations
* To determine the concordance of DNA and RNA alterations
* To determine the frequency of molecularly matched therapy
* To determine the feasibility of identifying mechanism(s) of acquired resistance with genomic profiling
* To determine the feasibility of molecularly matched therapy to acquired resistance alterations

Exploratory Objectives:

* To determine the feasibility of prioritizing targets with precision analytics
* To determine clinical outcomes in patients receiving molecularly matched therapy
* To determine the role of additional emerging diagnostic technologies

ELIGIBILITY:
Patient Eligibility:

Inclusion Criteria:

1. Male/female patients who are at least 18 years of age on the day of informed consent signing.
2. Patients must have a histologically documented diffuse large B-cell lymphoma requiring therapy.
3. Provision of written informed consent for the study.

Exclusion Criteria:

1. None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2027-05-12 (Estimated); Study Completion 2027-05-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who have genomic test results available in <=7 days | through study completion an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jason Westin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org